CLINICAL TRIAL: NCT02919657
Title: Genepro Gen2 Equivalency Study as Compared to Whey Isolate (1 Tablespoon of Genepro Gen2 and 30g Whey Isolate.
Brief Title: Absorption Comparison on Equivalency Value of Genepro Gen2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Musclegen Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Genepro Gen 2
Record Dates: First submitted 2016-09-19; First posted 2016-09-29 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Analysis, Event History; Absorption; Disorder, Protein
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genepro Gen2 Protein (Active Comparator): 1 tablespoon Serving of Genepro Gen2 Protein daily will be used in each subject.
  Intervention: Weekly blood draws will determine the effect on blood protein levels.
  Interventions: Dietary Supplement: Genepro Protein
- Whey Protein Isolate (Active Comparator): 30g Serving of Whey Isolate Protein will be used daily in each subject.
  Intervention: Weekly blood draws will determine the effect on blood protein levels.
  Interventions: Dietary Supplement: Whey Protein

INTERVENTIONS:
Dietary Supplement: Genepro Protein — weekly blood draws to measure blood protein levels
  Other Names: Genepro
  Arms: Genepro Gen2 Protein
Dietary Supplement: Whey Protein — weekly blood draws to measure blood protein levels
  Other Names: Whey Protein Isolate
  Arms: Whey Protein Isolate

SUMMARY:
Genepro Gen2 Absorption and Protein Value Clinical Trial.

DETAILED DESCRIPTION:
Objective: To prove the absorbability and usability of Genepro Gen2 Protein and compared to whey isolate. This study is intended to show the equivalent value of Genepro Gen2 as compared to whey protein isolate (1 tablespoon Genepro Gen2 compared to 30g serving of whey isolate)

Parameters: This study encompasses a 12-week program that follows 20 gastric bypass patients that have undergone weight loss surgery. We took a baseline blood analysis prior to the start of the study and subsequently we took weekly blood work to chart and register the findings. For this study we will only be doing the weekly analysis on blood protein levels by utilizing Spectrophotometry. The target blood protein range is 6.1-8.7 g/dL this test is administered while fasting.

Participants: 20 Post Op Gastric Bypass patients. 10 men, 10 women. All participants were between the ages of 30-46 years of age. All participants have been post operation from their weight loss surgery for a minimum of 3 months prior to the start of the study and no longer than 12 months at the start of the study.

Gathering Results: 10 subjects will receive Genepro Gen 2 protein (1 tablespoon serving) for the first 6 weeks of the study and for the last six weeks, they will receive 30g of Whey protein. In conjunction the other group of 10 subjects will receive 30g whey protein the first 6 weeks of the study and Genepro Gen2 protein the final six weeks. Weekly blood analysis will determine blood protein levels.

Diet: Diet guidelines limit the calories you consume while providing you with balanced meals to help prevent nutritional deficiencies and preserve your muscle tissue. Each patient tolerates suggested foods differently.

Daily calories should be between 600 to 700 for the duration of this study. Each subject is to follow a diet low in calories, fats and sweets. The goal for each subject is to consume a minimum of 65 to 75 grams of protein a day. High protein foods include eggs, meats, fish, seafood, tuna, poultry, tofu, milk, soy, cottage cheese, and yogurt. 30g of each daily intake of protein will be provided by a powdered protein supplement. Each subject will utilize a 30g serving of whey isolate for 6 weeks of their study and for the other 6 weeks the subject will use a single serving (1tablespoon) of Genepro Gen2 Protein.

Subject were given the following eating guidelines:

* Eat slowly and chew small bites of food thoroughly.
* Avoid rice, bread, raw vegetables, fresh fruits, and meats that are not easily chewed such as pork and steak. Ground meats are usually better tolerated.
* With soft and solid foods, take only three bites at one sitting, then wait a minimum of 20 minutes before eating more.
* Eat balanced meals with small portions.
* Avoid the use of drinking straws and carbonated beverages, chewing gum and ice because they can introduce too much air into your pouch and cause discomfort.
* Avoid sugar, sugar-containing foods and beverages, concentrated sweets, and fruit juices Alcoholic beverages will have a more profound effect and should be avoided or consumed with caution.

Exercise: Each subject is asked to exercise for 30 to 45 minutes a day, with cardio or aerobic activity three to five times a week. Initially, we recommend walking five minutes in the morning and five minutes in the late afternoon. As tolerated you should increase these intervals by five minutes until you are walking at least 15 minutes twice per day.

ELIGIBILITY:
* 20 Post Op Gastric Bypass patients.
* 10 men,
* 10 women.
* Minimum age 30
* Maximum age 46
* All participants have been post operation from their weight loss surgery for a minimum of 3 months prior to the start of the study and no longer than 12 months at the start of the study.

Exclusion Criteria:

* Any digestive distress disorder (IBS, Crones, etc).

Ages: 30 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Michael, RN, Principal Investigator — Musclegen Research, Inc.; Brian M Parks, PHD, Study Director — MedFit Rx, Inc.; Tony R Parks, BS, Principal Investigator — MedFit Rx, Inc.

IPD SHARING:
Plan to Share IPD: Yes
10 subjects will be administered genepro for the first 6 weeks of the study and whey protein the last 6 week. The other 10 subjects will be administered whey protein for the first 6 weeks of the study and Genepro Gen2 for the last 6 weeks. Weekly blood draws will be taken from each subject to analyze blood protein levels.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open call for bariatric patients via social media and direct mail marketing.
Groups:
- Genepro Gen2 Protein Then Whey Protein: 1 tablespoon Serving of Genepro Gen2 Protein daily will be used in each subject.
  30g Serving of Whey Isolate Protein will be used daily in each subject.
- Whey Protein Isolate Then Genepro Gen2 Protein: 30g Serving of Whey Isolate Protein will be used daily in each subject.
  1 tablespoon Serving of Genepro Gen2 Protein daily will be used in each subject.
Period: Overall Study
Arm/Group | Genepro Gen2 Protein Then Whey Protein | Whey Protein Isolate Then Genepro Gen2 Protein
Started | 10 (10 Participants) | 10 (10 Participants)
Completed | 10 (completed with the same initial 10 participants) | 10 (completed with the same initial 10 participants)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 Post Op Gastric Bypass patients. 10 men, 10 women. All participants were between the ages of 30-46 years of age. All participants have been post operation from their weight loss surgery for a minimum of 3 months prior to the start of the study and no longer than 12 months at the start of the study.
Groups:
- All Participants: All participants were given a baseline blood analysis
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20
Protein blood levels [Mean (Standard Deviation); unit: g/dl] — Population: Participants assessed separately for each sequence.
  g/dl
    Genepro Gen2 first: number analyzed (Participants) | 10
    Genepro Gen2 first | 7.1 (.4)
    Whey Isolate first: number analyzed (Participants) | 10
    Whey Isolate first | 6.9 (.4)
    All Participants | 7.0 (.4)

OUTCOME MEASURES:

1. Primary Outcome: Weekly Blood Draws to Measure Blood Protein Levels
Description: Each week the 20 participants will have blood drawn to measure their blood protein levels.
  Each participant was required to give blood weekly to determine the blood protein levels. The results show the average over each six week period of testing for each row. Each participant was examined to see if they achieved the average range as set fourth by the dieticians of greater than 6.1 and less than 8.7 within a 10% variable as acceptable.
  10 Participants will be given Genepro Gen2 for the first six weeks of the study and whey protein for the final 6.
  10 Participants will be given when protein for the first six weeks of the study and Genepro Gen2 for the final 6.
  These measurements will read in g/dl
Time Frame: 6 weeks per intervention
Measure: Mean (Standard Deviation); unit: grams per deciliter
Groups:
- Genepro Gen2 Protein: 1 tablespoon Serving of Genepro Gen2 Protein daily will be used in each subject.
  Intervention: Weekly blood draws will determine the effect on blood protein levels.
  Genepro Protein: weekly blood draws to measure blood protein levels
- Whey Protein Isolate: 30g Serving of Whey Isolate Protein will be used daily in each subject.
  Intervention: Weekly blood draws will determine the effect on blood protein levels.
  Whey Protein: weekly blood draws to measure blood protein levels
Arm/Group | Genepro Gen2 Protein | Whey Protein Isolate
Number analyzed (Participants) | 20 | 20
grams per deciliter
  Female Age 37 | 7.23 (.4) | 6.86 (.4)
  Male Age 34 | 7.43 (.7) | 7.21 (.3)
  Male Age 30 | 7.1 (.5) | 7.28 (.2)
  Female Age 32 | 7.16 (.3) | 6.95 (.1)
  Female Age 40 | 7.2 (.3) | 6.86 (.2)
  Male Age 40 | 7.11 (.8) | 6.08 (1.1)
  Male B Age 34 | 7.05 (.6) | 6.95 (.5)
  Female Age 34 | 6.6 (.2) | 6.46 (.3)
  Female B Age 37 | 6.55 (.2) | 6.65 (.2)
  Male Age 39 | 7.18 (1.1) | 6.88 (.3)
  Female Age 30 | 6.81 (.5) | 6.58 (.2)
  Male Age 46 | 6.81 (.5) | 6.58 (.2)
  Female Age 39 | 6.76 (.3) | 6.03 (.5)
  Male Age 36 | 6.81 (.5) | 6.48 (.2)
  Female B Age 32 | 6.88 (.6) | 6.26 (.4)
  Male Age 38 | 7.18 (.5) | 6.83 (.8)
  Female Age 36 | 6.73 (.9) | 6.31 (.4)
  Male C Age 34 | 7.13 (.4) | 7 (.4)
  Female B Age 36 | 6.13 (.8) | 6 (.8)
  Male Age 41 | 7 (.5) | 6.95 (.3)

ADVERSE EVENTS:
Description: No adverse events were monitored
Arm/Group | Genepro Gen2 Protein | Whey Protein Isolate
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other